CLINICAL TRIAL: NCT01244204
Title: Vitamin D Supplementations as Adjunct to Anti-tuberculosis Drugs in Mongolia
Brief Title: Role of Vitamin D in Innate Immunity to Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Ganmaa Davaasambuu, Assistant Professor of Medicine, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1K99HL089710-01A1 (NIH)
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Vitamin D Deficiency; Tuberculosis
Keywords: vitamin D deficiency; tuberculin sin test; immunity; tuberculosis
MeSH Terms: conditions — Vitamin D Deficiency; Tuberculosis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental)
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Daily dose of 800IU of vitamin D
  Arms: Vitamin D
Dietary Supplement: Placebo — Identically appearing capsules
  Arms: Placebo

SUMMARY:
The investigators proposed a pilot study preparatory to developing a randomized trial of vitamin D for the prevention of TB infection. The specific aims are presented below:

1. To recruit subjects, obtain consent, distribute vitamin D supplements to the children in the schools, obtain blood samples and transport them to the United States.
2. To test the hypothesis that daily vitamin D supplementation will increase plasma levels of 25(OH)D, and restore TLR-induced antimicrobial activity in monocytes/macrophages tested in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be children age 12 to 15 years inclusive in public school, located in Songino-Khairhan district, who are residents of Ulaanbaatar, and whose parents have given informed consent and who accent to participate in the study.

Exclusion Criteria:

* Individuals with pre-existing calcium, parathyroid conditions, or type I diabetes, sarcoidosis, or who require chronic diuretic therapy including calcium channel blockers, or who are cognitively impaired.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Serum vitamin D levels | 6 months
Tuberculin Skin Test conversion | 6 monhs

REFERENCES:
- [Derived] Yegorov S, Bromage S, Boldbaatar N, Ganmaa D. Effects of Vitamin D Supplementation and Seasonality on Circulating Cytokines in Adolescents: Analysis of Data From a Feasibility Trial in Mongolia. Front Nutr. 2019 Oct 23;6:166. doi: 10.3389/fnut.2019.00166. eCollection 2019. PMID 31709259
- [Derived] Ganmaa D, Giovannucci E, Bloom BR, Fawzi W, Burr W, Batbaatar D, Sumberzul N, Holick MF, Willett WC. Vitamin D, tuberculin skin test conversion, and latent tuberculosis in Mongolian school-age children: a randomized, double-blind, placebo-controlled feasibility trial. Am J Clin Nutr. 2012 Aug;96(2):391-6. doi: 10.3945/ajcn.112.034967. Epub 2012 Jul 3. PMID 22760564